CLINICAL TRIAL: NCT04910230
Title: Efficiency and Safety of Nicotinamide-based Supportive Therapy in Lymphopenia for Patients With COVID-19: A Randomized Clinical Trial
Brief Title: Nicotinamide-based Supportive Therapy in Lymphopenia for Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qiang Hu (Other)
Responsible Party: Sponsor-Investigator, Qiang Hu, Principal Investigator, Shenyang Northern Hospital
Organization: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N2020-12
Record Dates: First submitted 2021-05-24; First posted 2021-06-02 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Lymphopenia
Keywords: nicotinamide; COVID19; lymphopenia
MeSH Terms: conditions — COVID-19; Lymphopenia | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nicotinamide plus usual care (Experimental)
  Interventions: Drug: nicotinamide
- usual care (No Intervention)

INTERVENTIONS:
Drug: nicotinamide — In addition to usual care, the treatment group was given 500mg nicotinamide daily, divided into 5 doses
  Arms: nicotinamide plus usual care

SUMMARY:
The mechanism of peripheral blood lymphocyte decline in COVID-19 patients is not yet clear. However, one theory demonstrated that in the whole progression of COVID-19, the extensive activation of poly-ADP-ribose polymerase (PARP) may reduce the cellular NAD+ and dampen the adaptive immune system. So investigators presume that replenishing the NAD+ using nicotinamide as the precursor may improve the lymphocyte counts and boost the adaptive immune system. As a result, the study using nicotinamide as a kind of supportive therapy provide further evidence of their efficiency and safety in treating lymphopenia in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* the patients diagnosed as the common or severe cases of COVID-19
* aged 18-85
* the absolute lymphocyte counts below the normal value (<1.1-3.2×109/L)

Exclusion Criteria:

* the patients who are diagnosed as critically ill cases or participating in other clinical trials
* women who are pregnant or lactating
* ALT/AST > 5 times upper limit of normal (ULN), neutrophils counts < 0.5×109/L, platelets counts< 50×109/L
* patients diagnosed with rheumatoid immune-related diseases
* patients who take long-term oral anti-rejection drugs or immunomodulatory drugs
* hypersensitive reaction to nicotinamide or any auxiliary materials
* patients with active tuberculosis or combined with bacterial and fungal infections
* patients undergoing organ transplant
* patients with mental disorders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
changes in absolute lymphocyte counts | before and 48 hours after intervention
  the changes in absolute lymphocyte counts (*10^9/L) in before and 48 hours after treatment

SECONDARY OUTCOMES:
the death in hospital | before and 48 hours after intervention
  the rate of death in hospital (%)
the composite endpoint of aggravation | before and 48 hours after intervention
  the rate of composite endpoint of aggravation(%) , according to upgraded oxygen therapy, improvement of nursing level, and ward rounds of superior physicians for changes of conditions using the time to event principle. The upgraded oxygen therapy, improvement of nursing level, and ward rounds of superior physicians for changes of conditions would be combined to the composite endpoint in percentage (%). The upgraded oxygen therapy was defined as upgrading of ge neral high-volume oxygen intake from oxygen intake, ventilator using from high-volume oxygen intake or transference to intensive care unit from ventilator using.

CONTACTS AND LOCATIONS:
Overall Officials: Quan-Yu L Zhang, phD, Principal Investigator — Department of Cardiology, General Hospital of Northern Theater Command, Shenyang 110016, China
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Hu Q, Zhang QY, Peng CF, Ma Z, Han YL. Efficiency of nicotinamide-based supportive therapy in lymphopenia for patients with ordinary or severe COVID-19: A randomized controlled trial. Medicine (Baltimore). 2022 Oct 28;101(43):e31138. doi: 10.1097/MD.0000000000031138. PMID 36316932